CLINICAL TRIAL: NCT07230327
Title: Research on a New Disease Activity Assessment System for axSpA Based on Whole-body Magnetic Resonance Imaging Cohort
Brief Title: Whole Body MRI for Non-invasive Lesion Detection and Therapy Follow-up: Study With Patients With Radiographic axSpA and Non-radiographic axSpA
Acronym: NJSpAM
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Wenfeng Tan, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: SPA-JS
Record Dates: First submitted 2024-01-15; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Spondyloarthritis (SpA); Whole-body MRI (WBMRI)
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Procedure: Whole body MRI — These studies will be performed on a 3Tesla (T) MR system (Achieva, Philips Medical Systems) for all patients.

SUMMARY:
This study aims to further improve and expand the WB-MRI imaging evaluation cohort of axSpA patients to complete dynamic follow-up and condition assessment. Based on the WB-MRI features, the association of WB-MRI signs with disease activity, inflammation, and structural damage will be analyzed. At the same time, in-depth data mining was conducted and machine learning was used to construct a new axSpA disease activity assessment model based on WB-MRI data, and the accuracy and reliability of the model were clearly evaluated in the discovery cohort and validation cohort.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a common clinical chronic inflammatory joint disease with a high disability rate. Current assessment of axSpA disease activity mainly relies on patients' self-reported symptoms and signs, which has poor accuracy and reliability. At the same time, existing assessment methods fail to include some important disease characteristics of axSpA, such as active spinal inflammation and enthesitis. Therefore, there is an urgent need to establish a new axSpA disease activity assessment system.

With the development of imaging technology, whole-body MRI (WB-MRI) scanning technology is highly sensitive, can detect multiple parts at the same time, and can fuse multiple sequence images to make disease location and diagnosis more accurate. Currently, Much attention has been paid to it, but it has been less studied in axSpA.

This study established a disease activity assessment model based on WB-MRI imaging assessment, which will provide a new, effective and accurate method for axSpA disease assessment. At the same time, it will provide theoretical basis and practical basis for further understanding of the clinical characteristics of axSpA, the relationship between inflammation and structural damage.

ELIGIBILITY:
Inclusion Criteria:

Include newly referred patients if:

The onset of symptoms (back pain/arthritis/enthesitis) < 45 years

Undiagnosed disease with the following symptoms:

chronic back pain (duration of back pain more than 3 months) and/or peripheral arthritis (asymmetric arthritis/predominantly of the lower limbs) and/or enthesitis and/or dactylitis

Exclusion Criteria:

And diagnosed with non-radiographic or radiographic axial SpA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Exclusion Criteria:
  Unable to provide written consent Unable to undergo MRI examination Pregnancy Unable to read and/or write Chinese
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
WB-MRI imaging characteristics of patients with axSpA. | Two years
  Compare the correlation between WB-MRI changes and disease activity, disease progression and structural damage at baseline and after 2 years of follow-up.

SECONDARY OUTCOMES:
The correlation between WB-MRI changes and disease activities | Five yeas
  To elucidate the correlation between WB-MRI changes and inflammation, structural damage and disease activity in patients with axSpA.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Treitl KM, Ricke J, Baur-Melnyk A. Whole-body magnetic resonance imaging (WBMRI) versus whole-body computed tomography (WBCT) for myeloma imaging and staging. Skeletal Radiol. 2022 Jan;51(1):43-58. doi: 10.1007/s00256-021-03799-4. Epub 2021 May 24. PMID 34031705
- [Background] Hynes JP, Hughes N, Cunningham P, Kavanagh EC, Eustace SJ. Whole-body MRI of bone marrow: A review. J Magn Reson Imaging. 2019 Dec;50(6):1687-1701. doi: 10.1002/jmri.26759. Epub 2019 Apr 23. PMID 31016800
- [Background] Guo Z, Li B, Zhang Y, Kong C, Liu Y, Qu J, Zhan Y, Shen Z, Lei X. Peripheral enthesitis assessed by whole-body MRI in axial spondyloarthritis: Distribution and diagnostic value. Front Immunol. 2022 Aug 23;13:976800. doi: 10.3389/fimmu.2022.976800. eCollection 2022. PMID 36081521
- [Background] Poggenborg RP, Eshed I, Ostergaard M, Sorensen IJ, Moller JM, Madsen OR, Pedersen SJ. Enthesitis in patients with psoriatic arthritis, axial spondyloarthritis and healthy subjects assessed by 'head-to-toe' whole-body MRI and clinical examination. Ann Rheum Dis. 2015 May;74(5):823-9. doi: 10.1136/annrheumdis-2013-204239. Epub 2014 Jan 3. PMID 24389294
- [Background] Krabbe S, Ostergaard M, Eshed I, Sorensen IJ, Jensen B, Moller JM, Balding L, Madsen OR, Asmussen K, Eng G, Jorgensen NR, Pedersen SJ. Whole-body Magnetic Resonance Imaging in Axial Spondyloarthritis: Reduction of Sacroiliac, Spinal, and Entheseal Inflammation in a Placebo-controlled Trial of Adalimumab. J Rheumatol. 2018 May;45(5):621-629. doi: 10.3899/jrheum.170408. Epub 2018 Feb 15. PMID 29449506
- [Background] Karpitschka M, Godau-Kellner P, Kellner H, Horng A, Theisen D, Glaser C, Brandlhuber B, Reiser M, Weckbach S. Assessment of therapeutic response in ankylosing spondylitis patients undergoing anti-tumour necrosis factor therapy by whole-body magnetic resonance imaging. Eur Radiol. 2013 Jul;23(7):1773-84. doi: 10.1007/s00330-013-2794-1. Epub 2013 Mar 15. PMID 23494493
- [Background] Poggenborg RP, Pedersen SJ, Eshed I, Sorensen IJ, Moller JM, Madsen OR, Thomsen HS, Ostergaard M. Head-to-toe whole-body MRI in psoriatic arthritis, axial spondyloarthritis and healthy subjects: first steps towards global inflammation and damage scores of peripheral and axial joints. Rheumatology (Oxford). 2015 Jun;54(6):1039-49. doi: 10.1093/rheumatology/keu439. Epub 2014 Nov 26. PMID 25431482
- [Background] Weckbach S. Whole-body MRI for inflammatory arthritis and other multifocal rheumatoid diseases. Semin Musculoskelet Radiol. 2012 Nov;16(5):377-88. doi: 10.1055/s-0032-1329881. Epub 2012 Dec 4. PMID 23212873
- [Background] Althoff CE, Sieper J, Song IH, Haibel H, Weiss A, Diekhoff T, Rudwaleit M, Freundlich B, Hamm B, Hermann KG. Active inflammation and structural change in early active axial spondyloarthritis as detected by whole-body MRI. Ann Rheum Dis. 2013 Jun;72(6):967-73. doi: 10.1136/annrheumdis-2012-201545. Epub 2012 Jun 26. PMID 22736088
- [Background] Krabbe S, Eshed I, Sorensen IJ, Jensen B, Moller JM, Balding L, Madsen OR, Pedersen SJ, Ostergaard M. Whole-body Magnetic Resonance Imaging Inflammation in Peripheral Joints and Entheses in Axial Spondyloarthritis: Distribution and Changes during Adalimumab Treatment. J Rheumatol. 2020 Jan;47(1):50-58. doi: 10.3899/jrheum.181159. Epub 2019 Apr 1. PMID 30936290
- [Background] Weiss BG, Bachmann LM, Pfirrmann CW, Kissling RO, Zubler V. Whole Body Magnetic Resonance Imaging Features in Diffuse Idiopathic Skeletal Hyperostosis in Conjunction with Clinical Variables to Whole Body MRI and Clinical Variables in Ankylosing Spondylitis. J Rheumatol. 2016 Feb;43(2):335-42. doi: 10.3899/jrheum.150162. Epub 2015 Dec 15. PMID 26669910
- [Background] Althoff CE, Sieper J, Song IH, Weiss A, Diekhoff T, Haibel H, Hamm B, Hermann KG. Comparison of Clinical Examination versus Whole-body Magnetic Resonance Imaging of Enthesitis in Patients with Early Axial Spondyloarthritis during 3 Years of Continuous Etanercept Treatment. J Rheumatol. 2016 Mar;43(3):618-24. doi: 10.3899/jrheum.150659. Epub 2016 Feb 1. PMID 26834218